CLINICAL TRIAL: NCT02409563
Title: Effectiveness of Nasal Budesonide on Control of Airway Inflammation by Determining FeNO in Children With Allergic Rhinitis.
Brief Title: Nasal Budesonide Efficacy on Nasal FeNO in Children With Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Senior Researcher, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2/2013; ethics committee approval (Other: Verbale n. 2/2013)
Record Dates: First submitted 2013-02-07; First posted 2015-04-07 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Budesonide nasal (100 mcg bid) (Experimental): The study will be randomized, controlled parallel group. After 1 week of phase baseline screening (Visit 1), patients will be randomized (1:4) with the assignment of a code (B-200_da 01 to 08, B-100_ 01 to 31) (day 0, Visit 2) in 2 groups: N1 (n = 8) = Budesonide nasal spray 100 mcg, 2 v / d; Patients return to control after the 1st week (day 7, Visit 3), after the 2nd week (day 14, Visit 4) and one week after the end of the treatment period (day 21, Visit 5). It will give a tolerance of ± 3 days for the timing of planned visits. In the phase of follow-up, (3 days after the last dose of drug) will be recorded the occurrence of adverse effects (Adverse Event, EA)
  Interventions: Drug: Budesonide nasal spray (100 mcg bid)
- Budesonide nasal (50 mcg bid) (Experimental): The study will be randomized, controlled parallel group. After 1 week of phase baseline screening (Visit 1), patients will be randomized (1:4) with the assignment of a code (B-200_da 01 to 08, B-100_ 01 to 31) (day 0, Visit 2) in 2 groups: ; N2 (n = 31) = Budesonide nasal spray 50 mcg, 2 v / d. Patients return to control after the 1st week (day 7, Visit 3), after the 2nd week (day 14, Visit 4) and one week after the end of the treatment period (day 21, Visit 5). It will give a tolerance of ± 3 days for the timing of planned visits. In the phase of follow-up, (3 days after the last dose of drug) will be recorded the occurrence of adverse effects (Adverse Event, EA)
  Interventions: Drug: Budesonide nasal spray (50 mcg bid

INTERVENTIONS:
Drug: Budesonide nasal spray (100 mcg bid)
  Arms: Budesonide nasal (100 mcg bid)
Drug: Budesonide nasal spray (50 mcg bid
  Arms: Budesonide nasal (50 mcg bid)

SUMMARY:
In clinical trials for treatment of allergic rhinitis a significant reduction of the total symptom score compared to baseline has been demonstrated by using nasal budesonide.Previous results in adults show that the assessment and monitoring del nasal fractional exhaled nitric oxide (nFeNO) is useful in controlling inflammation of nasal allergic rhinitis.

Primary objective of this study is to evaluate efficacy of nasal budesonide (aqueous solution) on the nasal inflammation marker (nFeNO).

Secondary outcomes are the evaluation of: changes in total nasal symptom score (Total Symptom Score, T5SS), changes in cell counts in nasal lavage (LN) and the changes reported sleep quality (Pittsburgh Sleep Quality Index, PSQI).

ELIGIBILITY:
Inclusion Criteria:

* history of allergic rhinitis for at least 1 year
* children aged 6 - 14 years
* Total Symptom Score (T5SS) more than 6 in the last 4 days before the screening visit

Exclusion Criteria:

* signs of acute respiratory infection
* systemic immunological and metabolic disease
* major malformations of the upper airways
* topical or systemic therapy with antibiotics, antihistamines and corticosteroids in the 30 days prior to the study
* patient active smoker

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Nasal nitric oxide (nFeNO) | 21 days
  Assessment of the influence of nasal Budesonide (aqueous solution) on nasal FeNo (nFeNO) in children with allergic rhinitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy

REFERENCES:
- [Result] Meltzer EO. Clinical and antiinflammatory effects of intranasal budesonide aqueous pump spray in the treatment of perennial allergic rhinitis. Ann Allergy Asthma Immunol. 1998 Aug;81(2):128-34. doi: 10.1016/S1081-1206(10)62798-6. PMID 9723557
- [Result] Pedroletti C, Lundahl J, Alving K, Hedlin G. Effect of nasal steroid treatment on airway inflammation determined by exhaled nitric oxide in allergic schoolchildren with perennial rhinitis and asthma. Pediatr Allergy Immunol. 2008 May;19(3):219-26. doi: 10.1111/j.1399-3038.2007.00613.x. PMID 18399898
- [Result] Meltzer EO, Munafo DA, Chung W, Gopalan G, Varghese ST. Intranasal mometasone furoate therapy for allergic rhinitis symptoms and rhinitis-disturbed sleep. Ann Allergy Asthma Immunol. 2010 Jul;105(1):65-74. doi: 10.1016/j.anai.2010.04.020. PMID 20642206
- [Result] Bellodi S, Tosca MA, Pulvirenti G, Petecchia L, Serpero L, Silvestri M, Sabatini F, Battistini E, Rossi GA. Activity of budesonide on nasal neutrophilic inflammation and obstruction in children with recurrent upper airway infections. A preliminary investigation. Int J Pediatr Otorhinolaryngol. 2006 Mar;70(3):445-52. doi: 10.1016/j.ijporl.2005.07.015. Epub 2005 Sep 2. PMID 16140398
- [Result] Baraldi E, Azzolin NM, Carra S, Dario C, Marchesini L, Zacchello F. Effect of topical steroids on nasal nitric oxide production in children with perennial allergic rhinitis: a pilot study. Respir Med. 1998 Mar;92(3):558-61. doi: 10.1016/s0954-6111(98)90308-0. PMID 9692122